CLINICAL TRIAL: NCT00822796
Title: Thermogard™ Efficacy Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in obtaining surrogate consent on critically ill subjects.
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Timothy F. Haley, Division Surgeon, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I.2008.030; CIRO 2008235
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Hypothermia; Burns
Keywords: Hypothermia; Severe burns; Warming catheter; Thermogard™; Coagulopathy
MeSH Terms: conditions — Hypothermia; Burns; Hemostatic Disorders | interventions — Rewarming

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Burn patients with >20% TBSA burns scheduled to undergo debridement and grafting who will have placed the Thermogard™ central venous warming catheter by Alsius
  Interventions: Device: Thermogard™
- B (Active Comparator): Burn patients with >20% TBSA burns scheduled to undergo debridement and grafting who will have placed a central venous catheter as a part of their routine burn management
  Interventions: Device: Standard central venous catheter

INTERVENTIONS:
Device: Thermogard™ — Those who have a Thermogard™ central venous warming catheter placed prior to surgery
  Other Names: Rewarming
  Arms: A
Device: Standard central venous catheter — Those who have a standard central venous catheter placed prior to surgery
  Arms: B

SUMMARY:
The purpose of this study is to determine if the Thermogard™ central venous catheter can prevent hypothermia (defined as a core body temperature less then 36.0 °C) in severely burned patients who are undergoing surgery for debridement and grafting in the setting of reduced ambient room temperature.

DETAILED DESCRIPTION:
Hypothermia in the severely burned has been shown to disrupt coagulation, impair myocardial function, weaken the host immune response, delay wound healing and increase mortality.

Current methods available for preventing and reversing hypothermia include administering heated, humidified oxygen, infusing warmed intravenous fluids centrally, performing peritoneal dialysis with warmed fluid, undergoing extracorporeal blood warming with partial bypass, and markedly increasing the ambient room temperature. These methods are either limited in their effectiveness or are impractical and potentially dangerous. Furthermore, the practice of markedly increasing the ambient room temperature creates a hostile work environment for health care providers which may impact patient care.

The FDA has classified the Alsius Thermogard™ heat exchange catheter as a Class II devices under 21 C.F.R §§ 870.5900. It is used in various clinical applications for cooling patients but it has not been FDA-approved for use in warming burn patients. The Thermogard™ is an integrated electro-mechanical heater/cooler that consists of a temperature monitor, a temperature controller unit, a heat exchanger unit, and roller pump. It supplies temperature controlled sterile saline to the indwelling catheter that is placed percutaneously in the patient. The catheter can be placed in the femoral vein (larger catheter with three heat exchange balloons) or the subclavian or jugular vein (smaller catheter with two heat exchange balloons).

Sterile saline is warmed (to a maximum temperature of 38 °C) in the external device and then pumped through the balloons coaxially mounted on the catheter, enabling direct warming of the blood. The catheter contains a temperature probe enabling a 'closed loop' temperature control system; the temperature is set at the desired level (the range of the device is 28-38°C, which may vary according to the installed software), after which the device warms the patient to this level by increasing or decreasing the temperature of the circulating saline. The core temperature is then maintained at the desired level for as long as the attending physician deems necessary. The catheter also has two ports for central venous access, which can be used to administer medication and/or for blood sampling.

The purpose of this study is to determine if the Thermogard™ central venous catheter can significantly impact the heat stress environment of the operating room by allowing severely burned patients to undergo surgery for debridement and grafting at lower ambient operating room temperatures when compared to control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females ages 18-70 with greater than 20% TBSA burns requiring excision and grafting and in need of a central venous catheter per ICU admission criteria.
* Patient or patient's surrogate must be able to verbalize understanding and willingness to participate in the study and provide written informed consent

Exclusion Criteria:

* Pregnancy. All females admitted to the burn ICU undergo routine serum hCG to determine pregnancy status. Those found to be pregnant will be excluded from entry into the study
* Burn patients enrolled in recombinant Factor VII study due to the theoretical increased risk for clot formation
* Basic and advanced enlisted trainees
* Age greater than 70 years old due to increased mortality rate among those severely burned
* Conditions which make placement of a central venous catheters a greater than normal risk (vascular anomalies, previous vascular surgery, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Ambient room temperature | Intraoperative

SECONDARY OUTCOMES:
Compare the incidence, duration and severity of hypothermia, | Beginning of surgery to eight hours postoperative
Compare the need for perioperative blood and/or blood product transfusions as a function of the percent total body surface area (TBSA) excised and grafted during surgery | Beginning of surgery to eight hours postoperative
Compare the incidence of foreshortened surgery due to refractory hypothermia defined as a persistent core body temperature less than 35.0 °C. | Intraoperative
Compare the difference between skin/core body temperature and the ambient room temperature of those physicians and associate staff members providing care to burn patients in the operating room | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F. Haley, MD, Principal Investigator — Brooke Army Medical Center; Steven E. Wolf, MD, Study Director — US Army Institute of Surgical Research

REFERENCES:
- [Background] Jurkovich GJ, Greiser WB, Luterman A, Curreri PW. Hypothermia in trauma victims: an ominous predictor of survival. J Trauma. 1987 Sep;27(9):1019-24. PMID 3656464
- [Background] Robinson S, Katariya K, et al. Perioperative temperature management: Roundtable discussion identifies need to avoid hypothermia. Minutes from the Anesthesia Patient Safety Foundation. 11 June 2005; Louisville, KY
- [Background] Frank SM, Fleisher LA, Breslow MJ, Higgins MS, Olson KF, Kelly S, Beattie C. Perioperative maintenance of normothermia reduces the incidence of morbid cardiac events. A randomized clinical trial. JAMA. 1997 Apr 9;277(14):1127-34. PMID 9087467
- [Background] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Background] Doufas AG. Consequences of inadvertent perioperative hypothermia. Best Pract Res Clin Anaesthesiol. 2003 Dec;17(4):535-49. doi: 10.1016/s1521-6896(03)00052-1. PMID 14661656
- [Background] Weinberg AD. Hypothermia. Ann Emerg Med. 1993 Feb;22(2 Pt 2):370-7. doi: 10.1016/s0196-0644(05)80467-6. PMID 8434836
- [Background] Gore DC, Beaston J. Infusion of hot crystalloid during operative burn wound debridement. J Trauma. 1997 Jun;42(6):1112-5. doi: 10.1097/00005373-199706000-00022. PMID 9210551
- [Background] Soung LS, Swank L, Ing TS, Said RA, Goldman JW, Perez J, Geis WP. Treatment of accidental hypothermia with peritoneal dialysis. Can Med Assoc J. 1977 Dec 17;117(12):1415-6. No abstract available. PMID 589543
- [Background] Wong PS, Pugsley WB. Partial cardiopulmonary bypass for the treatment of profound accidental hypothermic circulatory collapse. J R Soc Med. 1992 Oct;85(10):640. doi: 10.1177/014107689208501021. No abstract available. PMID 1433050
- [Background] El-Gamal N, Elkassabany N, Frank SM, Amar R, Khabar HA, El-Rahmany HK, Okasha AS. Age-related thermoregulatory differences in a warm operating room environment (approximately 26 degrees C). Anesth Analg. 2000 Mar;90(3):694-8. doi: 10.1097/00000539-200003000-00034. PMID 10702459
- [Background] Hancock PA, Vasmatzidis I. Effects of heat stress on cognitive performance: the current state of knowledge. Int J Hyperthermia. 2003 May-Jun;19(3):355-72. doi: 10.1080/0265673021000054630. PMID 12745975
- [Background] Koenders S, Struijs A, et al, Feasibility of an intravenous warming device to rewarm cardiac surgery patients. NJCC 2004;8:34.
- [Background] Karabinis A, Mandila C, Koukoulitsios G, Dounis G, Tsoutsos D. Using an intravascular device to reverse refractory burn-associated hypothermia. Anaesth Intensive Care. 2008 Nov;36(6):918-9. No abstract available. PMID 19117092
- [Background] Willekes T, Naunheim R, Lasater M. A novel method of intravascular temperature modulation to treat severe hypothermia. Emerg Med J. 2006 Oct;23(10):e56. doi: 10.1136/emj.2006.035360. PMID 16988294
- [Background] Arthurs Z, Cuadrado D, Beekley A, Grathwohl K, Perkins J, Rush R, Sebesta J. The impact of hypothermia on trauma care at the 31st combat support hospital. Am J Surg. 2006 May;191(5):610-4. doi: 10.1016/j.amjsurg.2006.02.010. PMID 16647346